CLINICAL TRIAL: NCT03308396
Title: Single Arm Phase Ib/II Study of Durvalumab and Guadecitabine in Advanced Kidney Cancer: Big Ten Cancer Research Consortium BTCRC-GU16-043
Brief Title: Study of Durvalumab and Guadecitabine in Advanced Kidney Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ajjai Alva, MD (Other)
Collaborators: AstraZeneca (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Ajjai Alva, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GU16-043
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Advanced Kidney Cancer; Kidney Cancer; Clear Cell Renal Cell Carcinoma
Keywords: Durvalumab; Guadecitabine
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — guadecitabine; durvalumab

STUDY DESIGN:
Intervention Model Description: Phase Ib/II
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): This is a non-randomized, single arm, open label Phase Ib/II study.
  Phase Ib:
  Days 1-5
  Guadecitabine:
  * Dose 0: 60 mg/m^2
  * Dose -1: 45 mg/m^2
  Phase II:
  Days 1-5 Guadecitabine (at Ph II dose)
  Day 8 Durvalumab (1500 mg IV) Day 8 Durvalumab (1500 mg IV)
  Interventions: Drug: Guadecitabine; Drug: Durvalumab

INTERVENTIONS:
Drug: Guadecitabine — Days 1-5 Dose 0: 60 mg/m^2 Dose -1: 45 mg/m^2
  Other Names: SGI-110
Drug: Durvalumab — Day 8 Durvalumab (1500 mg IV)
  Other Names: MEDI4736

SUMMARY:
This is a single arm, multi-centre (via Big Ten Cancer Research Consortium) phase Ib/II study of patients treated with durvalumab 1500 mg IV q 4 weeks in combination with guadecitabine at the recommended phase 2 dose subcutaneously for 5 consecutive days. Eligible patients will have metastatic RCC with a clear cell component, ECOG performance status of 0-1, have received 0-1 prior therapy but no prior anti-PD-1/PD-L1/CTLA4 (Cohort 1, 36 subjects). Study treatment could potentially continue for up to 13 cycles (52 weeks).

DETAILED DESCRIPTION:
A total of up to 58 subjects will be enrolled on both phases.

Phase Ib: 6-12 subjects; enrolled into either Cohort 1 or 2. Phase II: 46 subjects; enrolled into either Cohort 1 or 2.

Cohort 1 (36 subjects): received 0-1 prior therapy and no prior anti-PD-1/PD-L1/CTLA4.

Cohort 2 (16 subjects): received up to 2 prior therapies, one of which must include an anti-PD-1/PD-L1 therapy to which they did not respond. Only one prior anti-PD-1/PD-L1 therapy is allowed.

Patients from Phase Ib treated at the eventual phase II dose will be combined with patients in Phase II in the efficacy analysis.

* Therapy will start with guadecitabine on days 1-5 of a 28-day cycle. Guadecitabine will be dosed subcutaneously on days 1-5 at either dose level 0 (60 mg/m2) or dose level -1 (45 mg/m2), based on the recommended phase II dose.
* Durvalumab will be started on day 8 of the 28-day cycle. Durvalumab will be administered intravenously at a flat dose of 1500mg every 28 days.
* Study treatment may continue for up to 13 cycles (52 weeks) in the absence of confirmed progression, intolerable toxicity, or withdrawal of consent.

Phase Ib Treatment Plan

* Dose limiting toxicities (DLTs) will be evaluated within the first cycle (i.e., within the first 28 days).
* Six patients will be enrolled at dose level 0. If 2 or fewer patients experience a dose limiting toxicity, the study will continue to the phase II portion at dose level 0.
* Alternately, if 3 or more patients have a dose limiting toxicity at dose level 0, 6 patients will be accrued at the lower dose (dose -1). If 2 or fewer patients experience a dose limiting toxicity, the study will continue to phase II at dose level -1.
* If 3 or more subjects experience a dose limiting toxicity at dose level -1, the treatment will be considered unsafe and the trial will be stopped. In this case, durvalumab and guadecitabine will be permanently discontinued and the subjects followed per protocol.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information.
* ECOG Performance Status 0-1 within 28 days prior to registration.
* Histological diagnosis of clear cell renal cell carcinoma (pure or mixed) with radiologic or histologic evidence of metastatic disease.
* At least 1 lesion, not previously irradiated that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have a short axis ≥ 15mm) with a computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements as per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) guidelines.
* For cohort 1, subjects may have received up to 1 and no more than 1 prior line of systemic therapy (not counting any neoadjuvant/adjuvant therapy) including anti-VEGF, VEGFR inhibitor, MET inhibitor or mTOR inhibitor for metastatic disease. They cannot have received any prior anti-PD-1/PD-L1/CTLA4 therapy including durvalumab.
* For cohort 2, subjects may have received up to 2 prior systemic therapies which should include 1 (and only 1) prior anti-PD-1/PD-L1 therapy but did not have an objective response to the prior anti-PD-1/Pd-L1 therapy. The treating investigator must document that the patient did not have an objective response to prior anti-PD-1/PD-L1 therapy. They may have received prior anti-CTLA4 therapy.
* Subjects may not have had radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* Prior cancer treatment must be completed at least 14 days prior to study registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤Grade 1 or baseline.
* Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 28 days prior to registration:

Hematological:

* White blood cell (WBC) ≥ 3 K/mm^3
* Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm^3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets (Plt) ≥ 100,000/mm^3

Renal:

* Calculated creatinine clearance ≥ 40 cc/min using the Cockcroft-Gault formula

Hepatic:

* Total Bilirubin ≤ 1.5 × upper limit of normal (ULN), except in cases of Gilbert's syndrome where the criteria will be ≤ 5 x ULN
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN

  * Females of childbearing potential must have a negative serum pregnancy test within 28 days prior to registration.
  * Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use at least 1 highly effective methods of contraception from the time of informed consent until 30 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
  * Life expectancy ≥ 12 weeks (in the opinion of the Investigator)
  * Body weight >30kg
  * Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Active infection requiring systemic therapy.
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry. Patients whose brain metastases have been treated may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration provided they show radiographic stability (defined as 1 brain image, obtained after treatment to the brain metastases). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable without the use of steroids for at least 14 days prior to the start of treatment.
* Pregnant or breastfeeding
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* Treatment with any investigational drug within 14 days prior to study registration.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]) within the last 3 years prior to study registration. The following are exceptions to this criterion: The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia.
  * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Subjects without active disease in the last 5 years may be included but only after consultation with the study physician.
  * Subjects with celiac disease controlled by diet alone.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca/ MedImmune staff and/or staff at the study site).
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Any concurrent chemotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g. hormone replacement therapy) is acceptable. Note: Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable (e.g., local surgery or radiotherapy).
* Major surgical procedure (as defined by the Investigator) within 28 days prior to study registration. Note: local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation that requires use of immunosuppressive agents.
* Uncontrolled intercurrent illness including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of leptomeningeal carcinomatosis.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study drug.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of study drug.
* Known allergy or hypersensitivity to study drugs or other humanized monoclonal antibodies.
* Patient ≤30kg in weight.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

  * Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose limiting toxicities will be assessed to determine if the trial is stopped before the Phase II portion. | 28 days/First cycle
  Number of patients with dose-limiting toxicity (DLT) of the combination of durvalumab and guadecitabine
Objective response rate | 1 year
  Objective response rate (complete response (CR) + partial response (PR)) by RECIST 1.1 in Cohort 1

SECONDARY OUTCOMES:
Phase II: Overall Survival (OS) | 2 years
  will be reported with 95% confidence intervals from the Kaplan-Meier estimates.
Phase II: Duration of Response (DoR) | 2 years
  will be assessed using Kaplan-Meier estimates including the 95% confidence band separately for cohort 1 and for cohort 2.
Phase II: Progression-free survival (PFS) | 2 years
  will be assessed using Kaplan-Meier estimates including the 95% confidence band separately for cohort 1 and for cohort 2.
Phase II: Clinical benefit rate (CBR) | 2 years
  reported as binomial proportions and corresponding 95% binomial confidence intervals separately for cohort 1 and cohort 2
Phase II: Complete response (CR) proportion | 2 years
  reported as binomial proportions and corresponding 95% binomial confidence intervals separately for cohort 1 and cohort 2
Phase II: Objective Response Rate (ORR) | 2 years
  reported as binomial proportions and corresponding 95% binomial confidence intervals separately for cohort 1 and cohort 2
Phase II: Assess Adverse Events | 2 years
  by CTCAE ver 4 including events of special interest such as immune mediated toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, M.D., Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - Univerisity of Illinois Cancer Center, Chicago, Illinois
  - University of Iowa Hosptials and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Penn State Cancer Institute, Hershey, Pennsylvania

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org